CLINICAL TRIAL: NCT03468010
Title: Adjuvant Chemotherapy Versus Observation After Radiation With Concurrent Cisplatin of Cervical Cancer (With Pelvic or Para-aortic Node Involvement) :A Phase 3 Prospective Multi-institutional Randomised Controlled Trial
Brief Title: A Trial Comparing Adjuvant Chemotherapy With Observation After Concurrent Chemoradiotherapy of Cervical Cancer (With Pelvic or Para-aortic Node Involvement)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Wei-jun Ye, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2017-105-01
Record Dates: First submitted 2018-03-10; First posted 2018-03-16 (Actual); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Cervical Cancer; Adjuvant Chemotherapy; Radiation; Lymph Node Metastases
MeSH Terms: conditions — Uterine Cervical Neoplasms; Lymphatic Metastasis | interventions — Chemoradiotherapy; TP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The control group (Group A) (Active Comparator): In Group A, observation is given after chemoradiation
  Interventions: Radiation: chemoradiation
- The experiment group (Group B) (Experimental): in Group B, three cycles of Paclitaxel, Cisplatin are administered after radiation with concurrent cisplatin. The regimen of additional adjuvant chemotherapy following radiation is Paclitaxel 135mg/m2 plus Cisplatin 60mg/m2 once 3 weeks.
  Interventions: Radiation: chemoradiation; Drug: Paclitaxel, Cisplatin

INTERVENTIONS:
Radiation: chemoradiation — radiation with concurrent ciplatin
Drug: Paclitaxel, Cisplatin — The regimen of additional adjuvant chemotherapy following radiation is Paclitaxel, Cisplatin once 3 weeks.
  Arms: The experiment group (Group B)

SUMMARY:
Cervical cancer with pelvic or para-aortic node involvement has a poor prognosis. Despite low-quality data, the routine practice to treat these patients is radiation with concurrent cisplatin. The aim of this study is to compare systemic chemotherapy with observation after radiation with concurrent cisplatin of cervical cancer ( with pelvic or para-aortic node involvement) for incidence of adverse events and local recurrence rate.

DETAILED DESCRIPTION:
1. Background Cervical Cancer is one of the most common malignant tumors of Chinese females. Women with evidence of para-aortic node involvement have a poor prognosis with a five-year survival rate of approximately 40 percent. Despite low-quality data, the routine practice to treat these patients is radiation with concurrent cisplatin. It is not clear whether systemic chemotherapy delivered following RT will obtain survival benefit.
2. Objective The aim of this study is to compare systemic chemotherapy with observation after radiation with concurrent cisplatin of cervical cancer ( with pelvic or para-aortic node involvement) for incidence of adverse events, 3y-PFS and 5y-OS, .
3. Patients

A patient will be enrolled when patient have:

1. Pathologically diagnosed cervical cancer;
2. pelvic or para-aortic lymph metastases, at least match one of following

   * CT or MRI scan shows pelvic or para-aortic node with a minimal axial diameter diameter ≥ 7mm in the largest plane
   * pelvic or para-aortic lymph node shows necrosis or extra capsular spread
   * PET/CT scan finds positive pelvic or para-aortic node lymph node
   * biopsy confirms lymph metastase
3. Stage IB1-IVA diseases (FIGO system ver. 2014) without treatment before;
4. Karnofsky Performance Scores ≥ 70;

4.Method

1. Randomization is performed to divide the patients into the control group (Group A) and the experimental group (Group B). In Group A, observation is given after radiation with concurrent cisplatin. But in Group B, three cycles of adjuvant chemotherapy ( Paclitaxel plus Cisplatin) are administered after radiation with concurrent cisplatin. The regimen of adjuvant chemotherapy following radiation is Paclitaxel 135mg/m2 plus Cisplatin 60mg/m2 once 3 weeks.The Grade 3/4 adverse events (CTCAE criteria ver. 4.03), the 3-year progression-free survival of the 2 groups, the 5-year overall survival of the 2 groups are compared.
2. In Group A and Group B, both the radiation method and the regimen of concurrent chemotherapy are the same.The gross tumor volume (GTVnd) is the lymph node lesion and given a dose of 60Gy. The clinical target volume (CTV) is according to the lymph drainage pathway and given a dose of 45Gy. The regimen of concurrent chemotherapy is Cisplatin 80mg/m2 once three weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically diagnosed cervical cancer;
2. pelvic or para-aortic lymph metastases, at least match one of following

   * CT or MRI scan shows pelvic or para-aortic node with a minimal axial diameter diameter ≥ 7mm in the largest plane
   * pelvic or para-aortic lymph node shows necrosis or extra capsular spread
   * PET/CT scan finds positive pelvic or para-aortic node lymph node
   * biopsy confirms lymph metastase
3. Stage IB1-IVA diseases (FIGO system ver. 2014) without treatment before;
4. Karnofsky Performance Scores ≥ 70;

Exclusion Criteria:

1. Patients with distant metastasis before or during radiotherapy
2. Severe dysfunction of heart, lung, liver, kidney or hematopoietic system
3. Severe neurological, mental or endocrine diseases
4. History of other malignancies
5. Those who are considered by the researchers unsuitable to participate -

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
3-year progression-free survival (3y-PFS) | 3 years after the date of adjuvant chemotherapy completion
  Percentage of patients in a treatment group who are alive without disease get worse for a 3-year period of follow-up after the date of adjuvant chemotherapy completion

SECONDARY OUTCOMES:
Incidence of grade 3/4 adverse event | Once a week during therapy, up to 5 years after the date of adjuvant chemotherapy completion
  Incidence of patients in a treatment group who manifest a specific adverse event (such as myelosuppression) of grade 3/4. Incidence is calculated for each adverse event respectively and severity is evaluated on basis of Common Terminology Criteria for Adverse Events (CTCAE) criteria ver. 4.03.

OTHER OUTCOMES:
5-year overall survival (5y-OS) | 5 years after the date of adjuvant chemotherapy completion
  Percentage of patients in a treatment group who are alive for a 5-year period of follow-up after the date of adjuvant chemotherapy completion

CONTACTS AND LOCATIONS:
Overall Officials: Wei-jun Ye, M.D, Principal Investigator — Sun Yat-sen University
Locations (8):
- China (8):
  - Sun Yat-sen University Affiliated Foshan Hospital, Foshan, Guangdong
  - Hospital of of Guangdong Armed Police Corps, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The First affiliated Hospital of Guangdong Pharmaceutical University, Guangzhou, Guangdong
  - Guangzhou First People's Hospital, Guanzhou, Guangdong
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Hainan General Hospital, Haikou, Hainan
  - Xinjiang Medical University Affiliated Tumor Hospital, Ürümqi, Xinjiang

IPD SHARING:
Plan to Share IPD: No